CLINICAL TRIAL: NCT03666000
Title: A Phase 1/1b, Open-label, Dose-escalation, Dose-expansion, Parallel Assignment Study to Evaluate Safety and Clinical Activity of PBCAR0191 (Azercabtagene Zapreleucel or "Azer-cel") in Subjects With Relapsed/Refractory (r/r) Non-Hodgkin Lymphoma (NHL) and r/r B-cell Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: Dose-escalation and Dose-expansion Study of Safety of Azer-cel (PBCAR0191) in Participants With Relapsed/Refractory (r/r) Non-Hodgkin Lymphoma (NHL) and r/r B-cell Acute Lymphoblastic Leukemia (B-ALL)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Imugene Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBCAR0191-01
Record Dates: First submitted 2018-08-20; First posted 2018-09-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Non-Hodgkin Lymphoma; B-cell Acute Lymphoblastic Leukemia; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; Cyclophosphamide; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1 Dose Escalation: Azer-cel Dose Level 1 (Experimental): Azer-cel, 3 x 10^5 CAR T cells per kilogram (kg) body weight.
  Route of Administration: Intravenous infusion
  Interventions: Biological: Azer-cel; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 1 Dose Escalation: Azer-cel Dose Level 2 (Experimental): Azer-cel, 1 x 10^6 CAR T cells per kg body weight.
  Route of Administration: Intravenous infusion
  Interventions: Biological: Azer-cel; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 1 Dose Escalation: Azer-cel Dose Level 3a (Experimental): Azer-cel, 3 x 10^6 CAR T cells per kg body weight.
  Route of Administration: Intravenous infusion
  Interventions: Biological: Azer-cel; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 1 Dose Escalation: Azer-cel Dose Level 4 (Experimental): Azer-cel, 6 x 10^6 CAR T cells per kg body weight as 2 administrations of 3 x 10^6 CAR T cells per kg body weight on Day 0 and Day 10.
  Route of Administration: Intravenous infusion
  Interventions: Biological: Azer-cel; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 1 Dose Escalation: Azer-cel Dose Level 4b (Experimental): Azer-cel, 500 x 10^6 CAR T cells (flat dose).
  Route of Administration: Intravenous infusion
  Interventions: Biological: Azer-cel; Drug: Fludarabine; Drug: Cyclophosphamide
- Phase 1B Dose Expansion: Azer-cel (Experimental): Azer-cel will be administered at a dose level established in Phase 1.
  Route of Administration: Intravenous infusion
  Interventions: Biological: Azer-cel; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: IL-2

INTERVENTIONS:
Biological: Azer-cel — Infusion of Allogeneic Anti-CD19 CAR T cells
  Other Names: Allogeneic Anti-CD19 CAR T cells; PBCAR0191
Drug: Fludarabine — Specified dose on specified days
Drug: Cyclophosphamide — Specified dose on specified days
Drug: IL-2 — Specified dose on specified days
  Arms: Phase 1B Dose Expansion: Azer-cel

SUMMARY:
This is a Phase 1/1b, nonrandomized, open-label, parallel assignment, dose-escalation, and dose-expansion study to evaluate the safety and clinical activity of azer-cel, an allogeneic anti-CD19 CAR T, in adults with r/r B ALL, r/r B-cell NHL and CLL/SLL.

DETAILED DESCRIPTION:
This is a multicenter, nonrandomized, open-label, parallel assignment, dose-escalation, and dose-expansion study to evaluate the safety and tolerability, find an appropriate dose to optimize safety and efficacy, and evaluate clinical activity of azer-cel in participants with relapsed/refractory (r/r) B-cell acute lymphoblastic leukemia (B-ALL), non-Hodgkin lymphoma (NHL), and chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL). Before initiating azer-cel, participants will be administered lymphodepletion (LD). At Day 0 of the Treatment Period, participants will receive an intravenous (IV) infusion of azer-cel potentially followed by interleukin-2 (IL-2). All participants will be monitored through D720 or progression. All participants who receive a dose of azer-cel will be asked to consent to a separate long-term follow-up (LTFU) study for up to 15 years after exiting this study.

ELIGIBILITY:
Key Inclusion Criteria

Criteria for B-ALL:

• Participant has confirmed unequivocal r/r CD19+ B-ALL.

Criteria for NHL and CLL/SLL:

• Participant has unequivocal aggressive CD19+ r/r B-cell NHL that is confirmed by tumor biopsy tissue from last relapse after CD19-directed therapy.

For Phase 1 Dose Escalation:

* Diffuse large B-cell lymphoma (DLBCL) including Richter's transformation
* Follicular lymphoma (FL) including Grade 3 or transformed FL
* High-grade B-cell lymphoma (HGBCL)
* Primary mediastinal lymphoma

For Phase 1b Dose Expansion (CAR T-relapsed cohort):

* DLBCL not otherwise specified (NOS)
* HGBCL
* DLBCL transformed from the following indolent lymphoma subtypes (FL, Marginal Zone lymphoma [MZL], and Waldenstrom's Macroglobulinemia [WM])
* Other large B-cell lymphoma (LBCL) subtypes may be enrolled with approval from the Medical Monitor.
* Participants previously treated with CD19-directed autologous CAR T therapies have received no more than 2 lines of therapy after administration of their previous CAR T product.
* For the expansion CAR T-relapsed cohort only: Participants must have received autologous CD19-directed CAR T therapy and demonstrated clinical response to the treatment at Day 28 or later, followed by relapse or progression.

For Phase 1b dose expansion (CAR T-naive cohort):

* DLBCL NOS
* DLBCL transformed from the following indolent lymphoma subtypes (FL, MZL, and WM)
* HGBCL
* FL (Grade 1-3a)
* MZL that is fluorodeoxyglucose (FDG)-avid on positron emission tomography (PET) scan
* WM
* CLL/SLL
* Primary central nervous system (CNS) lymphoma (PCNSL)
* Other LBCL subtypes may be enrolled with approval from the Medical Monitor.
* Participant must have received at least 1-2 prior lines of therapy, depending on histological subtype but no more than 7 systemic lines of anti-cancer therapy.

Criteria for both B-ALL, NHL, and CLL/SLL:

* Eastern Cooperative Oncology Group performance status score of 0 or 1.
* An estimated life expectancy of at least 12 weeks according to the investigator's judgment.
* Seronegative for human immunodeficiency virus antibody.
* Participant has adequate bone marrow, renal, hepatic, pulmonary, and cardiac function.

Key Exclusion Criteria

Criteria for B-ALL:

• Burkitt cell (L3 ALL) or mixed-lineage acute leukemia.

Criteria for NHL:

* Requirement for urgent therapy due to tumor mass effects such as bowel obstruction or blood vessel compression.
* Active hemolytic anemia.

Criteria for B-ALL and NHL:

* No active CNS disease, excluding PCNSL
* History of another primary malignancy
* Any form of primary immunodeficiency (for example, severe combined immunodeficiency disease).
* History of hepatitis B or hepatitis C currently receiving ongoing antiviral therapy.

Any known uncontrolled cardiovascular disease at the time of Screening that, in the investigator's opinion, renders the participant ineligible

* History of hypertension crisis or hypertensive encephalopathy within 3 months prior to Screening.
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Presence of a CNS disorder that, in the opinion of the investigator, renders the participant ineligible for treatment.
* History of concomitant genetic syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman-Diamond syndrome, or any other known bone marrow failure syndrome.
* Active uncontrolled autoimmune disease requiring active immunosuppression at the time of Screening (excluding participants needing steroids for physiologic replacement).
* Participant has received stem cell transplant within 90 days before Screening.
* Participant has active graft-versus-host disease (GvHD) symptoms.
* Participant has received a systemic biologic agent for treatment of the disease under study within 28 days of LD, other systemic anti-cancer therapy within 10 days or 5 half-lives (whichever is shorter) of LD, and no pulse steroid for disease control within 3 days of LD.
* Radiotherapy within 4 weeks before Screening.
* Presence of pleural/peritoneal/pericardial catheter, as well as permeant biliary and ureteral stents (does not apply to intravenous lines).
* Participant has received live vaccine within 4 weeks before Screening. Note: Non-live virus vaccines are not excluded.
* Participant has received CD19-directed therapy other than autologous CD19-directed CAR T therapy within 90 days of the anticipated start date of LD.

Additional criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Dose Escalation/Phase 1b Dose Expansion: Number of Participants with Azer-cel-related AEs Defined as Dose-limiting Toxicities (DLTs) | Up to Day 720
Phase 1b Dose Expansion: Objective Response Rate (ORR) B-ALL | Up to Day 720
  ORR for participants with B-ALL will be assessed by National Comprehensive Cancer Network (NCCN) 2017 criteria.
Phase 1b Dose Expansion: ORR NHL | Up to Day 720
  ORR for participants with NHL will be assessed by Lugano classification, International Workgroup on Chronic Lymphocytic Leukemia (iwCLL) 2018 guidelines, International Primary Central Nervous System Lymphoma Collaborative Group (IPCG) criteria, and International Workshop on Waldenstrom's Macroglobulinemia (IWWM)-11 criteria.

SECONDARY OUTCOMES:
Phase 1 Dose Escalation: ORR | Up to Day 720
  * B-ALL: NCCN 2017 criteria
  * NHL: Lugano classification
Complete Response (CR) Rate | Up to day 720
  * B-ALL: NCCN 2017 criteria
  * NHL: Lugano classification
Duration of Response (DoR) | Up to day 720
  - Defined as the duration (days) from initial response to disease progression or death.
Progression-free survival (PFS) | Up to day 720
  - Defined as the duration (days) from Day 0 to disease progression or death.
Overall survival (OS) | Up to day 720
  - Defined as the duration (days) from Day 0 to death.
Time to next treatment (TNT) | Up to day 720
  - Defined as the duration (days) from Day 0 to institution of next systemic therapy.
Number of Participants with AEs | Up to day 720
  - Defined as all AEs of clinical significance captured on study and specific reporting of DLTs, treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interests (AESIs), and AEs related to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John Byon, MD, PhD, Study Chair — Imugene Limited
Locations (23):
- United States (18):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - City of Hope, Duarte, California
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - Northside Hospital Cancer Institute, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute (Wayne State University), Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Weill Cornell Medical College - NY Presbyterian Hospital, New York, New York
  - Columbia University Irving Medical Center/New York Presbyterian Hospital, New York, New York
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Lifespan Cancer Institute at Rhode Island Hospital, Providence, Rhode Island
  - Baylor University Medical Center, Dallas, Texas
  - MD Anderson, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Barwon Health - Andrew Love Cancer Centre, Geelong, Victoria

IPD SHARING:
Plan to Share IPD: No